CLINICAL TRIAL: NCT07335978
Title: The Role of Chair Exercise and Intergenerational Activities in Older Adults With Physico-Cognitive Decline Syndrome: An Investigation of Frailty and Serum Mature Brain-Dervied Neurotrophic Factor Level
Brief Title: Chair Exercise and Intergenerational Activities in Older Adults With Physio-Cognitive Decline Syndrome
Acronym: PCDS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atma Jaya Catholic University of Indonesia (Other)
Responsible Party: Principal Investigator, Agnes Rensa, Princial Investigator, Atma Jaya Catholic University of Indonesia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 25-06-0948
Record Dates: First submitted 2026-01-02; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cognitive Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Nutritional education + 12 weeks structured chair-based exercise (PEROSI protocol, progressive frequency from 1 to 3 sessions/week, 60 minutes/session, supervised online) followed sequentially by 4 weeks SHP-based intergenerational activities (8 sessions, 2x/week, 45 minutes/session, paired 1:1 elderly-child using AMIR educational materials at selected orphanages).
  Interventions: Behavioral: Intervention 1
- Control Arm (No Intervention)

INTERVENTIONS:
Behavioral: Intervention 1 — Nutritional education + 12 weeks structured chair-based exercise (PEROSI protocol, progressive frequency from 1 to 3 sessions/week, 60 minutes/session, supervised online) followed sequentially by 4 weeks SHP-based intergenerational activities (8 sessions, 2x/week, 45 minutes/session, paired 1:1 elderly-child using AMIR educational materials at selected orphanages).
  Arms: Intervention Arm

SUMMARY:
The goal of this clinical trial is to investigate the effects of chair exercise followed by intergenerational activity in frailty syndrome and changes in serum mBDN levels among older adults with Physio-Cognitive Decline Syndrome (PCDS), as a novel approach integrating physical and social intervention with biomolecular assessments

In older adults with PCDS

1. Does A 16-week program of chair exercise followed by intergenerational activity improve handgrip strength (HGS), gait speed, MoCA-Ina scores, and health-related quality of life?
2. Does a 16-week program of chair exercise followed by an intergenerational activity increase serum mBDNF level?
3. Are serum mBDNF levels associated with MoCA-Ina scores, gait speed, and handgrip strength?

Intervention Group

Participants will undergo a 12-week structured chair exercise program, conducted with a trained exercise instructor and supervised by a physician for vital sign monitoring during each session. The frequency of sessions will increase progressively:

* Weeks 1-2: once weekly
* Weeks 3-6: twice weekly
* Week 7-12: three times weekly

Additional activities include (intervention and control group):

* Weeks 1 and 11: teleconference session on nutrition and physical exercise supported by electronic flyers (e-flyers).
* Weeks 3, 5, 7, 11, and 13: distribution of e-flyers on elderly nutrition and the muscle-brain axis.

Additional Activity (intervention group)

- Weeks 13-16: intergenerational activities at an orphanage with children aged >5 years

Assessments (intervention and control group):

* Week 1: serum mBDNF and HbA1c measurement
* Week 12 and 16: physical assessments (body weight, height, handgrip strength, gait speed, MoCA-Ina, and IADL) and serum mBDNF measurement.

Control Group:

The participant will receive general health education on performing physical exercise 1-3 times per week throughout week 1-16

DETAILED DESCRIPTION:
Population aging in Indonesia has led to a growing proportion of older adults experiencing functional and cognitive decline. Physio-cognitive decline syndrome (PCDS), defined as the coexistence of reduced physical performance (such as slow gait speed or weak handgrip strength) and mild cognitive impairment without disability or dementia, is considered an early and reversible stage that increases the risk of frailty, disability, and poor quality of life.

Chair exercise provides a safe and feasible intervention for older adults, with proven benefits in muscle strength, balance, and neurocognitive function, partly mediated through increased levels of brain-derived neurotrophic factor (BDNF). In parallel, an intergenerational activity involving direct interaction between older and younger individuals has shown promise in improving psychosocial well-being and cognitive outcomes.

This study integrates chair exercise with intergenerational activities to target the multidimensional nature of PCDS. Outcomes will focus on frailty status and changes in serum mature brain-derived neurotrophic factor (mBDNF) to establish a multimodal, culturally adapted strategy to support healthy aging in Indonesian older adults.

ELIGIBILITY:
* Aged 60-75 years
* Meet diagnostic criteria for physio-cognitive decline syndrome (PCDS): gait speed <1.0 m/s and/or hand grip strength <28 kg (men) or <18 kg (women), and MoCA-Ina score 22-26
* Instrumental Activities of Daily Living (IADL) score >5
* Able to understand and follow instructions adequately
* Willing to participate and provide written informed consent

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-02-06 (Estimated); Study Completion 2026-02-13 (Estimated)

PRIMARY OUTCOMES:
Frailty Syndrome Status | From enrollment to the end of treatment at 12 weeks
  • Change in frailty syndrome status (assessed using Cardiovascular Health Study criteria: score 0 robust, 1-2 pre-frail, ≥3 frail) from baseline to week 16.
serum mature brain-derived neurotrophic factor (mBDNF) | from baseline to week 16
  Change in serum mature brain-derived neurotrophic factor (mBDNF) levels (measured by ELISA) from baseline to week 16.

SECONDARY OUTCOMES:
Hand grip strength | from baseline to week 16
  Change in hand grip strength (in kilogram; dominant hand, best of 3 trials using hand dynamometer) from baseline to week 16.
Gait Speed Test | baseline to week 16
  Change in gait speed (m/s; average of 2 trials over 6-meter walk test) from baseline to week 16.
Cognitive Function | from baseline to week 16
  Change in cognitive function (MoCA-Ina total score, range 0-30)
health-related quality of life (SF-12 questionnaire) | from baseline to week 16
  Change in health-related quality of life (SF-12 questionnaire)
serum mBDNF levels | baseline to week 16
  Correlations between changes in serum mBDNF levels and changes in MoCA-Ina score, hand grip strength, and gait speed.

OTHER OUTCOMES:
Adherence to exercise sessions | from baseline to week 12
  Adherence to exercise sessions
Intergenerational activities | from weeks 13 to weeks 16
  Adherence to intergenerational activities (attendance logs)
Physical Activity Scale for the Elderly, PASE | from baseline to week 16
  Physical activity level (Physical Activity Scale for the Elderly, PASE).
Depressive Symptoms | from baseline to week 16
  Questionnaire of Geriatric Depression Scale-15, GDS-15
Loneliness | From baseline to weeks 16
  Questionnaire of De Jong Gierveld Loneliness Scale, Indonesian version
Quality of Life Additional Domains | from baseline to week 16
  Questionnaire of Quality of life additional domains (EQ-5D-5L)
Charison Comorbidity Index (CCI) | baseline
  Questionnaire of Charison Comorbidity Index (CCI)

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic Church of St. Anthony of Padua, Bidaracina, GKI Depok, Catholic Church of St. Anna, Catholic Chrusch St. Aloysius Gonzaga, Jakarta, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT07335978/Prot_SAP_000.pdf